CLINICAL TRIAL: NCT03479970
Title: Rehabilitation of Social Cognition in Subjects With Traumatic Brain Injury. Efficiency of a Computer Rehabilitation Treatment
Brief Title: Rehabilitation of Social Cognition in Subjects With Traumatic Brain Injury
Acronym: SOCCER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Guttmann (Other)
Responsible Party: Principal Investigator, Pablo Rodriguez, Principal Investigator, Institut Guttmann
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017257
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Cognition Disorders
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNPT + Social Cognition (Experimental): Experimental Group: will undertake a rehabilitation treatment integrated by a set of tasks aimed at working attention, memory and executive functions together with a computerized treatment for the rehabilitation of the Social Cognition. The treatment will be carried out through the cognitive telerehabilitation platform Guttmann, NeuroPersonalTrainer® (GNPT).
  The treatment will consist of the carrying out of 24 treatment sessions
  Interventions: Other: GNPT+ Social Cognition
- GNPT (only N-SC measures) (Active Comparator): Control Group: will only conduct a cognitive rehabilitation treatment through the cognitive telerehabilitation platform Guttmann, NeuroPersonalTrainer® (GNPT) focused on attention, memory and executive functions.
  Interventions: Other: GNPT

INTERVENTIONS:
Other: GNPT+ Social Cognition — Aplication of a computer based treatment focused on attention, memory, executive functions and social cognition.
  Arms: GNPT + Social Cognition
Other: GNPT — It's a computeritzed program of cognitive telerehabilitation
  Arms: GNPT (only N-SC measures)

SUMMARY:
In the present study the investigators aim to analyze the performance in a battery of social cognition tests of subjects with traumatic brain injury.

On the other hand, the effectiveness of a computerized rehabilitation program designed to improve these deficits will be tested, as well as the relationship between social cognition and executive functioning.

DETAILED DESCRIPTION:
The ability of the individual to know how to adopt the perspective of the other or be able to interpret and correctly identify their emotions, is essential for their proper development in society. The term Social Cognition would be the construct that would encompass these cognitive processes.

People who have suffered a moderate or severe traumatic brain injury usually show, as reflected in the existing literature, an alteration in the functioning of Social Cognition, leading to problematic or inappropriate behaviors. These deficits have devastating consequences, at a personal, family and economic / labor level.

There is an important debate regarding the independence of the Social Cognition construct from the rest of cognitive functions and in particular with respect to executive functions, probably due to the overlapping of the neuroanatomical structures related to each of these functions.

In the present study a clinical trial will be conducted with a sample of 30 patients admitted to the Guttmann Institute Neurorehabilitation Hospital who have suffered a moderate or severe TBI.

Patients will be divided into two groups depending on whether they receive cognitive rehabilitation treatment focused on attention, memory and executive functions (Control Group) or if, in addition to this treatment, the computerized treatment module for the rehabilitation of CS is also applied. (Experimental Group). Both types of treatment would be carried out using the cognitive telerehabilitation platform Guttmann, NeuroPersonalTrainer® (GNPT).

The purpose of this study is to analyze the altered dimensions in the Social Cognition construct after having suffered a traumatic brain injury and to test the effectiveness of a computerized rehabilitation treatment designed for neuropsychologists with the aim of stimulating the relearning of these skills.

In the same way it is tried to establish and to clarify the existing relation between the construct of the social cognition and other cognitive functions as they can be the executive functions

ELIGIBILITY:
Inclusion Criteria:

* Age at the time of the TBI equal to or greater than 18 years.
* Evolution time between the TBI and the beginning of the participation in the study less than 6 months.
* Find out from the Post-Traumatic Amnesia Phase, evaluated through the Galveston Orientation and Amnesia Test (GOAT) scale: it is considered that the patient is out of PTA if he obtains scores greater than 75 in two consecutive administrations.
* Cognitive impairment through the neuropsychological scan battery that is administered by clinical protocol.

Exclusion Criteria:

* Alteration of the language that compromises the complete application of the neuropsychological exploration battery.
* Psychiatric history or neurological involvement prior to TBI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-01-02 (Estimated); Study Completion 2022-01-02 (Estimated)

PRIMARY OUTCOMES:
International Affect Picture System (IAPS) | 1 day
  Designed to provide a standardized set of pictures for studying emotion and attention. This subtest has a puntuation range from 0 to 25, where higher values are considered to be a better outcome.
Pictures of facial Affect (POFA) | 1 day
  It is an assessment test of the ability to identify basic emotions in facial. This subtest has a puntuation range from 0 to 65, where higher values are considered to be a better outcome. expressions
The Moving Shapes Paradigm | 1 day
  Evaluation of the interaction between two triangles based on low level. This subtest has a puntuation range from 0 to 12, where higher values are considered to be a better outcome. inferences
Reading The Mind in the Eyes Test (RMET) | 1 day
  Advanced test of theory of mind. The subject must identify emotions in the eyes of photographed people. This subtest has a puntuation range from 0 to 36, where higher values are considered to be a better outcome.
Social Decision Making Task The Social Decision Making Task (SDMT) | 1 day
  Pseudo online test of catch and throw where the participant is required to use social feedback.

SECONDARY OUTCOMES:
Conners Continuous Performance Test (CPT-II) | 1 day
  To improve performance in sustained attention after receiving experimental intervention. Puntuation range from 0 to 100. The correct puntuation ranges from 40 to 60.
Rey Auditory Verbal Learning Test (RAVLT) | 1 day
  To improve performance in short-term, long-term and recognition. This test has puntuation range from 0 to 75.
Spanish phonemic fluency test- PMR | 1 day
  To improve performance in phonemic fluency after receiving experimental intervention. This subtest has a puntuation range from 0 to 100, where higher values are considered to be a better outcome.
Digit Span forward Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in span of immediate verbal recall after receiving experimental intervention. This subtest has a puntuation range from 2 to 9, where higher values are considered to be a better outcome.
Digit Span backward Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in working memory after receiving experimental intervention. This subtest has a puntuation range from 2 to 8, where higher values are considered to be a better outcome.
Letter-Number Sequencing Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in working memory after receiving experimental intervention. This subtest has a puntation range from 1 to 21, where higher values are considered to be a better outcome.
Digit Symbol-Coding Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in speed of processing. This subtest has a puntuation range from 1 to 133, where higher values are considered to be a better outcome.
Block Design Subtest from the Wechsler Adult Intelligence Scale (WAIS-III) | 1 day
  To improve performance in visuoconstruction and planning. This subtest has a puntuation range from 1 to 68, where higher values are considered to be a better outcome.
Stroop Color and Word test (Stroop Test) | 1 day
  To improve performance in inhibitory control. This subtest has a puntuation range from 1 to 100, where higher values are considered to be a better outcome.
Trail Making Test A (TMT-A) | 1 day
  To improve performance in visual attention. This subtest has a puntuation range from 1 to 999 seconds, where higher values are considered to be a worst outcome.
Trail Making Test B (TMT-B) | 1 day
  To improve performance in task-switching. This subtest has a puntuation range from 1 to 999 seconds, where higher values are considered to be a worst outcome.
Wisconsin Card Sorting Test (WCST) | 1 day
  To improve performance in cognitive flexibility. This subtest has a puntuation range from 1 to 6 categories, where higher values are considered to be a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Rodríguez, Principal Investigator — Institut Guttmann
Locations (1):
- Hospital de Neurorehabilitació Institut Guttmann, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Rodriguez-Rajo P, Garcia-Rudolph A, Sanchez-Carrion R, Aparicio-Lopez C, Ensenat-Cantallops A, Garcia-Molina A. Computerized social cognitive training in the subacute phase after traumatic brain injury: A quasi-randomized controlled trial. Appl Neuropsychol Adult. 2024 Jul-Aug;31(4):540-553. doi: 10.1080/23279095.2022.2042693. Epub 2022 Feb 23. PMID 35196474